CLINICAL TRIAL: NCT00601744
Title: Social-Psychological Aspects of Survivorship in Cancer Patients After Orbital Exenteration: Issues Stemming From Alterations of Normal Facial Appearance
Brief Title: Social-Psychological Aspects of Orbital Exenteration
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0584
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Eye Cancer
Keywords: Orbital Exenteration; Eye Cancer; Social-Psychological Aspects; Quality of Life; Questionnaire; Facial Appearance; Survey; Interview
MeSH Terms: conditions — Eye Neoplasms; Facies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: Diagnosis of orbital or head and neck cancer and a history of orbital exenteration.
  Interventions: Behavioral: Audio-Taped Interview; Behavioral: Questionnaire
- Family Member/Friend: Family member or close friend of a patient with a diagnosis of orbital or head and neck cancer and a history of orbital exenteration.
  Interventions: Behavioral: Audio-Taped Interview

INTERVENTIONS:
Behavioral: Audio-Taped Interview — Meeting with a research staff member either in person or by phone, lasting 2 to 2 1/2 hours
  Arm 1: Questions about emotional well-being, appearance, coping ability with the cancer, and the types of social relations and support available (such as relationships with friends and family)
  Arm 2: Questions regarding if and how social relations may have been affected by his/her cancer experiences after the orbital exenteration.
  Other Names: Survey; Questionnaire
Behavioral: Questionnaire — 5-10 minute questionnaire to be completed after the interview.
  Other Names: Survey
  Groups: Patient

SUMMARY:
The goal of this research study is to learn about the social and emotional factors that may affect the quality of life of patients with cancer of the eye or eye area who have had their facial appearance changed due to an orbital exenteration.

DETAILED DESCRIPTION:
Family Members:

Study Interview:

If you agree to take part in this study, you will meet with a research staff member (preferably in person, or else by phone) for an interview. During the interview, you will be asked questions about your demographic information (such as your age, education level, and marital status). You will be asked about your family member's medical history, emotional well-being, appearance, and the types of social relations and support in his/her life (such as relationships with friends and family).

You will also be asked if and how these social relations may have been affected by his/her cancer experiences after the orbital exenteration. The interview should take about 2 to 2 1/2 hours. It will be audio-taped, and the interviewer will be taking notes. Your responses in the interview will not be shared with the patient.

Additional Information:

If your interview responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive mental health screening.

Length of Study Participation:

After the interview, your participation in this study will be over.

This is an investigational study.

Up to 40 people (20 patients and 20 family members) will take part in this study. All will be enrolled at MD Anderson.

Patients:

Study Interview:

If you agree to take part in this study, a research staff member will schedule you for an interview. During the interview, you will be asked questions about your demographic information (such as your age, education level, and marital status) and medical history. You will also be asked about your emotional well-being, how you feel about your appearance, how you are coping with the cancer, and the types of social relations and support you have in your life (such as relationships with friends and family). The interview should take about 2 to 2 1/2 hours. It will be audio-taped, and the interviewer will be taking notes.

Additional Information:

Your responses in the interview will not be shared with your doctor. If you feel you need a doctor's opinion about anything that is asked about in the questionnaire (such as mental or emotional difficulties), please contact your doctor.

If your interview responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive mental health screening.

Interview for Family Members:

For each eligible patient who agrees to take part in this study, one family member must also agree to participate. Researchers will ask you for a family member whom researchers can contact by phone to ask if he or she would agree to take part in this study. Your family member's participation would involve being interviewed about his or her opinions of the same questions that you were asked about in your interview. If your family member agrees, his or her interview will be scheduled. If that family member does not agree to take part, another family member may take part in his or her place. If no family members agree to take part, your interview will not be scheduled and you will not be enrolled on the study.

Length of Study Participation:

After you complete the interview, your participation in this study will be over.

This is an investigational study.

Up to 40 people (20 patients and 20 family members) will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older (for both patient & family member).
2. Must be able to communicate in a meaningful manner with the investigators (for both patient & family member).
3. Must be able to provide written/oral informed consent to participate (for both patient & family member).
4. A diagnosis of orbital or head and neck cancer and a history of orbital exenteration (for patient only). A family member or close friend of a patient with a diagnosis of orbital or head and neck cancer and a history of orbital exenteration (for family member only).
5. Must have obvious facial appearance change in the orbital area due to cancer treatment (for patient only). A family member or close friend of a patient with obvious facial appearance change in the orbital area due to cancer treatment (for family member only).
6. Must have a family member willing to participate in a separate interview (for patient only). Must be willing to participate in a separate interview (for both patient & family member).
7. Must be English speaking (for both patient & family member).

Exclusion Criteria:

1. Significant pre-existing facial disfigurement from a congenital defect or other disease or injury (for patient only).
2. Has recurrence of cancer and currently under treatment (for patient only).
3. Diagnosis of a serious mental disorder involving psychotic processes (such as formal thought disorder and schizophrenia) documented in medical record or otherwise apparent (for both patient & family member).
4. A foreign national (an individual who does not normally reside in the United States). These patients are excluded due to the confounding variables that cultural differences and language barriers may introduce (for both patient & family member).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient diagnosis of orbital or head and neck cancer and a history of orbital exenteration. Family member or close friend of a patient with a diagnosis of orbital or head and neck cancer and a history of orbital exenteration.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
List of physical adaptation and social-psychological issues cancer patients who survive and suffer from changes in normal facial appearance as a result of orbital exenteration | Participants evaluated at one time point (Interview - Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Bita Esmaeli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org